CLINICAL TRIAL: NCT02021487
Title: Pilot Study Prok-Idm: Interest of Dosage of Prokinecitine in Acute Myocardial Infarction
Brief Title: Prokinecitine in Acute Myocardial Infarction
Acronym: Prok-Idm
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5515
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: ST Elevatation Myocardial Infarction (STEMI)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to investigate the presence of a substance in the blood called prokinecitine, which is released by the heart when a heart attack occurs. Several venous blood samples at the arm are withdrawn at admission, H6, H12, H24, H48 and H72 in order to measure the concentration of this substance in the blood. The usefulness of this new blood marker is going to be determsined to seek if it would be of help to better diagnose or estimate the gravity of heart infarction after a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute St elevation myocardial infarction of less than 6 hours
* Age>18 y/o

Exclusion Criteria:

* Previous myocardial infarction
* LBB, RBB
* Renal Insuffiency MDRD<30 mL/min
* Patient with Pace-Maker or ICD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute St elevation myocardial infarction of less than 6 hours
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Infarct size by MRI necrotic myocardial mass | 7 days
  Infarct size by MRI necrotic myocardial mass

CONTACTS AND LOCATIONS:
Overall Officials: Patrick OHLMANN, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, France